CLINICAL TRIAL: NCT00887770
Title: A Single-centre, Double-blind, Double-dummy, Randomised, Placebo-controlled, Four-period Crossover Study to Assess the Effect of Single Oral Doses of AZD5672 (600 mg and 150 mg) on QT/QTc Interval, Compared to Placebo, Using Moxifloxacin (Avelox®) as a Positive Control, in Healthy Male Volunteers
Brief Title: A Study to Investigate the Potential for AZD5672 to Affect the Electrical Conduction Pathways in the Heart
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: D1710C00006; Eudract No. 2009-009940-22
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2009-07-16 (Estimated); Status verified 2009-07

CONDITIONS: Rheumatoid Arthritis
Keywords: QTcF; Crossover; ICH E14; QT/QTc prolongation; Moxifloxacin; QT/QTc Interval
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — N-(1-(3-(3,5-difluorophenyl)-3-(4-methanesulfonylphenyl)propyl)piperidin-4-yl)-N-ethyl-2-(4-methanesulfonylphenyl)acetamide; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): 600mg AZD5672 + Moxifloxacin placebo
  Interventions: Drug: AZD5672; Drug: placebo
- B (Experimental): 100mg AZD5672 + Moxifloxacin placebo
  Interventions: Drug: AZD5672; Drug: placebo
- C (Active Comparator): AZD5672 placebo + Moxifloxacin 400mg
  Interventions: Drug: Moxifloxacin; Drug: placebo
- D (Placebo Comparator): AZD5672 placebo + Moxifloxacin placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AZD5672 — 12 x 50mg tablet, oral, single dose
  Arms: A
Drug: Moxifloxacin — 1 x 400mg capsule, oral, single dose
  Other Names: Avelox
  Arms: C
Drug: placebo — 12 x matched to AZD5672 50 mg tablet
  Arms: C; D
Drug: AZD5672 — 3 x 50mg tablet, oral. single dose
  Arms: B
Drug: placebo — 9 x matched to AZD5672 50mg tablet
  Arms: B
Drug: placebo — 1 x matched to Moxifloxacin capsule
  Arms: A; B; D

SUMMARY:
This study is being performed to investigate the potential for AZD5672 to affect the electrical conduction pathways in the heart. AZD5672 will be compared against a drug (moxifloxacin - a licensed antibiotic) known to have a detectable but safe change on the electrical conduction of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18 and 30 kg/m2 and a minimum weight of 50kg.
* Non-smoker

Exclusion Criteria:

* Marked QTc prolongation at baseline e.g. repeated demonstration of QTc interval >450ms or marked shortening of QTcF <350ms
* Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of the QTc Interval changes
* Use of concomitant medications that prolong QT/QTc interval

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2009-04; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Evaluate time-matched QTcF intervals of single dose AZD5672 600mg compared to placebo. | Up to 24 hours postdose

SECONDARY OUTCOMES:
Evaluate time-matched QTcF Intervals of single dose AZD5672 150mg compared to placebo. | Up to 24 hours postdose
To evaluate the change in time matched ECG parameters (QTcB, QTcX, RR, PR and QRS) of single dose AZD5672 600mg and 150mg compared to placebo | Up to 24 hours postdose
To further evaluate the safety and tolerability of single dose AZD5672 600mg and 150mg | Adverse events assessed throughout the whole study. Safety monitoring (BP, safety blood samples and ECG) conducted frequently throughout study and up to 72 hours post dose on treatment visits.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Layton, Study Director — AstraZeneca R&D, Alderley Park, UK; Darren Wilbraham, Principal Investigator — Guys Drug Research Unit, Newcomen St, London
Locations (1):
- Research Site, London, United Kingdom